CLINICAL TRIAL: NCT01649869
Title: A Phase II Randomized and Controlled Investigation of Six Weeks of Oral Valganciclovir Therapy in Infants and Children With Congenital Cytomegalovirus Infection and Hearing Loss
Brief Title: Valganciclovir Therapy in Infants and Children With Congenital CMV Infection and Hearing Loss
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11-0069
Record Dates: First submitted 2012-07-20; First posted 2012-07-25 (Estimated); Results first posted 2021-06-02 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2018-03-22

CONDITIONS: Cytomegalovirus Infection
Keywords: CMV; Cytomegalovirus; Hearing Loss; Infants; Valganciclovir
MeSH Terms: conditions — Cytomegalovirus Infections; Hearing Loss | interventions — Valganciclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Active Comparator): 27 Children between 1 month and 3 years of age (up to 4th birthday) with sensoneural hearing loss and documented CMV infection will receive valganciclovir HCl 16.0 mg/kg orally twice a day for 6 weeks
  Interventions: Drug: Valganciclovir
- Placebo (Placebo Comparator): 27 Children between 1 month and 3 years of age (up to 4th birthday) with sensoneural hearing loss and documented CMV infection will receive placebo orally twice a day for 6 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Placebo — Simple Syrup as 60-90% sucrose in purified water: given orally twice a day for 6 weeks
  Arms: Placebo
Drug: Valganciclovir — Valcyte (valganciclovir hydrochloride) 50 mg of valganciclovir free base per 1 mL, oral solution: given at 16.0 mg/kg, twice a day for 6 weeks.
  Arms: Active

SUMMARY:
This is an international, multi-center, double-blind, placebo-controlled evaluation valganciclovir treatment for up to 54 children (up to 4 years of age) with virologically-confirmed congenital CMV infection and hearing loss. Subject participation will be over a six-month period and study subjects will be stratified according to age. The primary objective is to assess whether a six-week course of oral valganciclovir can stabilize the hearing of children with congenital CMV infection who present with hearing loss.

DETAILED DESCRIPTION:
Congenital cytomegalovirus (CMV) infection is the most frequent known viral cause of mental retardation, and is the leading non-genetic cause of sensorineural hearing loss in many countries including the United States. This is a Phase II international, multi-center, double-blind, placebo-controlled evaluation of 6 weeks of oral valganciclovir treatment or 6 weeks of placebo for fifty-four male and female infants/toddlers 1 month through 3 years of age (up to 4 years of age) with virologically-confirmed congenital CMV infection and hearing loss. Patient who are between 1 month and 4 years of age and who have SNHL (Sensorineural Hearing Loss) and are eligible for enrollment. The expected study duration is 3.5 years from enrollment of first study subject. The primary objective is to assess whether a six week course of oral valganciclovir can stabilize the hearing of children with congenital CMV infection who present with hearing loss. The secondary objective is to define the following responses as a function of systemic exposure to ganciclovir (active metabolite of valganciclovir): CMV viral load in blood; CMV viral load in urine; and CMV viral load in saliva. Also, to define the safety and tolerability of valganciclovir in enrolled subjects. The tertiary objective is to define the pharmacokinetics of ganciclovir (metabolite) following administration of valganciclovir (prodrug) in enrolled subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent from parent(s) or legal guardian(s)
2. Sensorineural hearing loss (>/= 21dB in one or both ears, documented within 12 weeks prior to study entry)
3. Children from 1 month through 3 years of age (up to the 4th birthday)

Exclusion Criteria:

1. Imminent demise
2. Profound sensorineural hearing loss (> 90dB) in both ears
3. Patients receiving other antiviral agents or immune globulin
4. Gastrointestinal abnormality which might preclude absorption of an oral medication (e.g., a history of necrotizing enterocolitis)
5. Documented renal insufficiency, as noted by a creatinine clearance < 10 mL/min/1.73m2 at time of study enrollment
6. Breastfeeding from mother who is receiving ganciclovir, valganciclovir, foscarnet, cidofovir, or maribavir
7. Infants known to be born to women who are HIV positive (but HIV testing is not required for study entry).
8. Current receipt of other investigational drugs
9. Previous receipt of ganciclovir or valganciclovir
10. Known hypersensitivity to ganciclovir, valganciclovir, or components of the product
11. Inability to attend follow-up hearing and clinical assessments
12. Infants with Auditory neuropathy/dyssynchrony.
13. Children with another known etiology for SNHL (e.g. connexin 26, syndrome or metabolic disorder associated with SNHL, inner ear malformation and widened vestibular aqueducts, meningitis).

Exclusion of each of these conditions is not required for trial enrollment.

Ages: 1 Month to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2015-02-24 (Actual); Primary Completion 2019-12-24 (Actual); Study Completion 2019-12-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- United States (9):
  - Children's of Alabama Child Health Research Unit (CHRU), Birmingham, Alabama
  - Children's National Medical Center - Sheikh Zayed Campus - Infectious Disease, Washington D.C., District of Columbia
  - Washington University School of Medicine in St. Louis - Center for Clinical Studies, St Louis, Missouri
  - Steven and Alexandra Cohen Childrens Medical Center of New York - New Hyde Park - Infectious Disease, Manhasset, New York
  - University of Rochester Medical Center, Rochester, New York
  - Carolinas Medical Center - Pediatrics - Infectious Diseases, Charlotte, North Carolina
  - Nationwide Children's Hospital - Neonatology - Center for Perinatal Research, Columbus, Ohio
  - Rhode Island Hospital - Pediatrics, Providence, Rhode Island
  - Texas Medical Center - Texas Children's Hospital, Houston, Texas
- United Kingdom (9):
  - Bristol Royal Hospital for Children - Paediatric Immunology, Bristol, Bristol, City of
  - Saint George's Hospital - Pediatric Infectious Diseases, London, London, City of
  - Great Ormond Street Hospital - Infectious Diseases, London, London, City of
  - Birmingham Heartlands Hospital, Birmingham
  - Pennine Acute Hospitals NHS Trust, North Manchester General Hospital - Children's and Adolescent Services, Crumpsall
  - John Radcliffe Hospital - Children's Hospital - Paediatric Infectious Disease and Immunology, Headington, Oxford
  - The Great North Children's Hospital - Paediatric Immunology, Newcastle upon Tyne
  - Sheffield Children's Hospital - Immunology, Sheffield
  - Southampton Children's Hospital - Allergy, Immunology and Infection, Southampton, Hampshire

REFERENCES:
- [Derived] Kimberlin DW, Aban I, Peri K, Nishikawa JK, Bernatoniene J, Emonts M, Klein N, Bamford A, DeBiasi RL, Faust SN, Jones CE, McMaster P, Caserta M, Ahmed A, Sharland M, Demmler-Harrison G, Hackett S, Sanchez PJ, Shackley F, Kelly D, Dennehy PH, Storch GA, Whitley RJ, Griffiths P; Collaborative Antiviral Study Group (CASG). Oral Valganciclovir Initiated Beyond 1 Month of Age as Treatment of Sensorineural Hearing Loss Caused by Congenital Cytomegalovirus Infection: A Randomized Clinical Trial. J Pediatr. 2024 May;268:113934. doi: 10.1016/j.jpeds.2024.113934. Epub 2024 Feb 2. PMID 38309519

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For this study, subjects were enrolled once they signed the informed consent form (ICF). It was not until after hearing loss was confirmed by audiology testing and confirmation of congenital CMV by dried blood spot that a subject was randomized and started on study drug. This reduced protocol enrollment from 54 to 35.
Period: Overall Study
Arm/Group | Placebo | Active
Started | 18 | 17
Completed | 16 | 16
Not Completed | 2 | 1
Not completed — Family member illness | 1 | 0
Not completed — Required treatment outside protocol | 1 | 0
Not completed — Severe hearing loss borderline eligible | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Active | Total
Number analyzed (Participants) | 18 | 17 | 35
Age, Continuous [Median (Standard Deviation); unit: MONTHS] | 19.5 (13.1) | 17.8 (15.8) | 18.7 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 10 | 11 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 17 | 15 | 32
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 15 | 12 | 27
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 4 | 11
  United Kingdom | 11 | 13 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Ears That Had (1) Improved Hearing or no Change in Hearing (2) Worsened Hearing.
Description: A single, independent study audiologist who is masked (blinded) to treatment assignment will assess the audiology test battery for each subject and assign the classifications of normal hearing, mild hearing loss, moderate hearing loss, or severe hearing loss based upon their hearing thresholds (in decibels). The classifications will be assigned by ear (one for the left ear and one for the right ear), giving "total ear" classifications. At the analyses stage, the "best ear" classification for the subject at that study visit will be determined; for example, if a subject had mild hearing loss in their left ear and severe hearing loss in their right ear, then the "best ear" classification will be mild hearing loss. Not both ears are evaluable for all subjects. In some subjects, only one ear is evaluable.
Time Frame: Day 1 through Day 180
Measure: Number; unit: Ears
Units Other Than Participants: Ears
Arm/Group | Placebo | Active
Number analyzed (Participants) | 16 | 15
Number analyzed (Ears) | 28 | 26
Ears
  Improve + no change | 27 | 20
  Worsened | 1 | 6
Statistical Analysis 1: Comparison: Placebo vs Active; Test type: Superiority; p = 0.0859, Generalized linear model; Generalized linear model for binary outcome based on generalized estimating equations

2. Secondary Outcome: Number of Best Ear That Had (1) Improved Hearing or no Change in Hearing (2) Worsened Hearing [ex. Improved+ no Change (Normal to Normal) Versus Other].
Description: A single, independent study audiologist who is masked (blinded) to treatment assignment will assess the audiology test battery for each subject and assign the classifications of normal hearing, mild hearing loss, moderate hearing loss, or severe hearing loss based upon their hearing thresholds (in decibels). The classifications will be assigned by ear (one for the left ear and one for the right ear), giving "total ear" classifications. At the analyses stage, the "best ear" classification for the subject at that study visit will be determined; for example, if a subject had mild hearing loss in their left ear and severe hearing loss in their right ear, then the "best ear" classification will be mild hearing loss. For this outcome, we combine the improved hearing and no change for the special case only of normal to normal. Other category include worsened and no change from (1) mild to mild hearing loss, (2) moderate to moderate hearing loss, or (3) severe to severe hearing loss.
Time Frame: Day 1 through Day 180
Measure: Number; unit: Participants
Arm/Group | Placebo | Active
Number analyzed (Participants) | 15 | 12
Participants
  Improved + normal to normal | 9 | 6
  No change abnormal or worsened | 6 | 6
Statistical Analysis 1: Comparison: Placebo vs Active; Test type: Superiority; p = 0.7068, Fisher Exact

3. Secondary Outcome: Change in Best Ear Hearing Assessments [Improved Versus Other] Between Baseline and Study Month 6.
Description: A single, independent study audiologist who is masked (blinded) to treatment assignment will assess the audiology test battery for each subject and assign the classifications of normal hearing, mild hearing loss, moderate hearing loss, or severe hearing loss based upon their hearing thresholds (in decibels). The classifications will be assigned by ear (one for the left ear and one for the right ear), giving "total ear" classifications. At the analyses stage, the "best ear" classification for the subject at that study visit will be determined; for example, if a subject had mild hearing loss in their left ear and severe hearing loss in their right ear, then the "best ear" classification will be mild hearing loss.
Time Frame: Day 1 through Day 180
Measure: Number; unit: Participants
Arm/Group | Placebo | Active
Number analyzed (Participants) | 15 | 12
Participants
  Improved | 0 | 0
  No change or worsened | 15 | 12
Statistical Analysis 1: Comparison: Placebo vs Active; Test type: Superiority; p = 1, Fisher Exact

4. Secondary Outcome: Change in Best Ear Hearing Assessments [Worse + no Change (Abnormal to Abnormal) Versus Other] Between Baseline and Study Month 6.
Description: as for outcome 3
Time Frame: Day 1 through Day 180
Measure: Number; unit: Participants
Arm/Group | Placebo | Active
Number analyzed (Participants) | 15 | 12
Participants
  No change abnormal to abnormal + worsened | 6 | 6
  Improved + normal to normal | 9 | 6
Statistical Analysis 1: Comparison: Placebo vs Active; Test type: Superiority; p = 0.7068, Fisher Exact

5. Secondary Outcome: Change in Best Ear Hearing Assessments [Worse Versus Other] Between Baseline and Study Month 6.
Description: as for outcome 3
Time Frame: Day 1 through Day 180
Measure: Number; unit: Participants
Arm/Group | Placebo | Active
Number analyzed (Participants) | 15 | 12
Participants
  Worsened | 0 | 3
  Other | 15 | 9
Statistical Analysis 1: Comparison: Placebo vs Active; Test type: Superiority; p = 0.0752, Fisher Exact

6. Secondary Outcome: Change in Total Ear Hearing Assessments [Improved Versus Other] Between Baseline and Study Month 6.
Description: as for outcome 3
Time Frame: Day 1 through Day 180
Measure: Number; unit: Ears
Units Other Than Participants: Ears
Arm/Group | Placebo | Active
Number analyzed (Participants) | 16 | 15
Number analyzed (Ears) | 28 | 26
Ears
  Improved | 0 | 0
  Other | 28 | 26

7. Secondary Outcome: Change in Total Ear Hearing Assessments [Worse+ no Change (Abnormal to Abnormal) Versus Other] Between Baseline and Study Month 6.
Description: as for outcome 3
Time Frame: Day 1 through Day 180
Measure: Number; unit: Ears
Units Other Than Participants: Ears
Arm/Group | Placebo | Active
Number analyzed (Participants) | 16 | 15
Number analyzed (Ears) | 28 | 26
Ears
  worse + no change (abnormal to abnormal) | 19 | 20
  Other | 9 | 6
Statistical Analysis 1: Comparison: Placebo vs Active; Test type: Superiority; p = 0.4823, Generalized linear model; Generalized linear model for binary outcome using generalized estimating equations

8. Secondary Outcome: Change in Total Ear Hearing Assessments [Worse Versus Other] Between Baseline and Study Month 6.
Description: as for outcome 3
Time Frame: Day 1 through Day 180
Measure: Number; unit: Ears
Units Other Than Participants: Ears
Arm/Group | Placebo | Active
Number analyzed (Participants) | 16 | 15
Number analyzed (Ears) | 28 | 26
Ears
  Worsened | 1 | 6
  Other | 27 | 20
Statistical Analysis 1: Comparison: Placebo vs Active; Test type: Superiority; p = 0.0859, Generalized linear model; Generalized linear model for binary outcome using generalized estimating equations

9. Secondary Outcome: Association of Change in Viral Load (Blood) With Change in Total Ear Hearing at 6 Months
Description: Analysis of actual viral load was done using log base 10 transformation. Undetectable viral load value was replaced by a value of 10. A summary measure of the viral load over time considers all time points available by calculating the average area under the curve (AUC) (trapezoidal rule) applied to the log base 10 viral load. Average is based on the maximum period of time with viral load data for a given subject. The average or standardize AUC units is therefore the original AUC units of log 10 copies/ml*days divided by days in study which equals log 10 copies/ml.
Time Frame: At 6 months
Population: Analysis was stratified by hearing outcome--total analyzed is the sum of the number analyzed for 2 rows below
Measure: Mean (Standard Deviation); unit: log 10 copies/ml
Units Other Than Participants: Ears
Groups:
- Randomized Group: Randomized children between 1 month and 3 years of age (up to 4th birthday) with sensoneural hearing loss and documented CMV infection will receive placebo orally twice a day for 6 weeks
Arm/Group | Randomized Group
Number analyzed (Participants) | 31
Number analyzed (Ears) | 54
log 10 copies/ml
  Improved + normal to normal: number analyzed (Ears) | 15
  Improved + normal to normal | 1.396 (0.542)
  No change abnormal + worsened: number analyzed (Ears) | 39
  No change abnormal + worsened | 1.326 (0.566)
Statistical Analysis 1: Comparison: Randomized Group; Test type: Other — Association of binary outcome and continuous outcome; p = 0.8212, Generalized linear model; For binary outcome using generalized estimating equations

10. Secondary Outcome: Association of Change in Viral Load (Saliva) With Change in Total Ear Hearing at 6 Months
Description: Analysis of actual viral load was done using log base 10 transformation. Undetectable viral load value was replaced by a value of 10. A summary measure of the viral load over time considers all time points available by calculating the average area under the curve (AUC) (trapezoidal rule) applied to the log base 10 viral load. Average is based on the maximum period of time with viral load data for a given subject. The average or standardize AUC units is therefore the original AUC units or log 10 copies/ml*days divided by days in study which equals log 10 copies/ml.
Time Frame: At 6 months
Population: Analysis stratified by hearing outcome--total analyzed is the sum of the number analyzed for 2 rows belos
Measure: Mean (Standard Deviation); unit: log 10 copies/ml
Units Other Than Participants: Ears
Arm/Group | Randomized Group
Number analyzed (Participants) | 31
Number analyzed (Ears) | 54
log 10 copies/ml
  Improved + normal to normal: number analyzed (Ears) | 15
  Improved + normal to normal | 2.447 (1.715)
  No change abnormal + worsened: number analyzed (Ears) | 39
  No change abnormal + worsened | 2.290 (1.349)
Statistical Analysis 1: Comparison: Randomized Group; Test type: Other — Association of binary outcome and continuous outcome and continuous outcome; p = 0.8356, Generalized linear model; Generalized linear model for binary outcome using generalized estimating equations

11. Secondary Outcome: Association of Change in Viral Load (Urine) With Change in Total Ear Hearing at 6 Months
Description: as for outcome 9
Time Frame: At 6 months
Population: Analysis stratified by hearing outcome--total analyzed is the sum of the number analyzed for 2 rows below
Measure: Mean (Standard Deviation); unit: log 10 copies/ml
Units Other Than Participants: Ears
Arm/Group | Randomized Group
Number analyzed (Participants) | 29
Number analyzed (Ears) | 50
log 10 copies/ml
  Improved + normal to normal: number analyzed (Ears) | 15
  Improved + normal to normal | 3.562 (1.139)
  No change abnormal + worsened: number analyzed (Ears) | 35
  No change abnormal + worsened | 3.583 (1.370)
Statistical Analysis 1: Comparison: Randomized Group; Test type: Other — Association of binary outcome and continuous outcome; p = 0.7961, Generalized linear model; Generalized linear model for binary outcome using generalized estimating equations

12. Secondary Outcome: Association of Change in Viral Load (Blood) With Change in Best Ear Hearing at 6 Months
Description: as for outcome 9
Time Frame: At 6 months
Population: Analysis stratified by hearing outcome--total analyzed is the sum of the number analyzed for 2 rows below
Measure: Mean (Standard Deviation); unit: log 10 copies/ml
Arm/Group | Randomized Group
Number analyzed (Participants) | 27
log 10 copies/ml
  Improved + normal to normal: number analyzed (Participants) | 15
  Improved + normal to normal | 1.396 (0.542)
  No change abnormal + worsened: number analyzed (Participants) | 12
  No change abnormal + worsened | 1.359 (0.668)
Statistical Analysis 1: Comparison: Randomized Group; Test type: Other — Association of binary outcome and continuous outcome; p = 0.8675, Generalized linear model; Generalized linear model for binary outcome

13. Secondary Outcome: Association of Change in Viral Load (Saliva) With Change in Best Ear Hearing at 6 Months
Description: as for outcome 9
Time Frame: At 6 months
Population: Analysis stratified by hearing outcome--total analyzed is the sum of the number analyzed for 2 rows below
Measure: Mean (Standard Deviation); unit: log 10 copies/ml
Arm/Group | Randomized Group
Number analyzed (Participants) | 27
log 10 copies/ml
  Improved + normal to normal: number analyzed (Participants) | 15
  Improved + normal to normal | 2.447 (1.715)
  No change abnormal + worsened: number analyzed (Participants) | 12
  No change abnormal + worsened | 2.423 (1.484)
Statistical Analysis 1: Comparison: Randomized Group; Test type: Other — Association of binary outcome and continuous outcome; p = 0.9682, Generalized linear model; Generalized linear model for binary outcome

14. Secondary Outcome: Association of Change in Viral Load (Urine) With Change in Best Ear Hearing at 6 Months
Description: as for outcome 9
Time Frame: At 6 months
Population: Analysis stratified by hearing outcome--total analyzed is the sum of the number of analyzed for 2 rows below
Measure: Mean (Standard Deviation); unit: log 10 copies/ml
Arm/Group | Randomized Group
Number analyzed (Participants) | 25
log 10 copies/ml
  Improved + normal to normal: number analyzed (Participants) | 15
  Improved + normal to normal | 3.562 (1.139)
  No change abnormal + worsened: number analyzed (Participants) | 10
  No change abnormal + worsened | 3.831 (1.570)
Statistical Analysis 1: Comparison: Randomized Group; Test type: Other — Association of binary outcome and continuous outcome; p = 0.6063, Generalized linear model; Generalized linear model for binary outcome

15. Secondary Outcome: Detection of Viruria (Urine) by PCR Six Weeks After Trial Entry
Description: Each subject either has positive or negative PCR results. Virus is detected if the PCR is positive.
Time Frame: At 6 weeks (Day 42)
Measure: Number; unit: Participants
Arm/Group | Placebo | Active
Number analyzed (Participants) | 12 | 12
Participants
  Positive | 11 | 1
  Negative | 1 | 11
Statistical Analysis 1: Comparison: Placebo vs Active; Test type: Superiority; p = 0.0001, Fisher Exact

16. Secondary Outcome: Detection of Viruria (Urine) by PCR Six Month After Trial Entry
Description: Each subject either has positive or negative PCR results. Virus is detected if the PCR is positive.
Time Frame: At 6 months
Measure: Number; unit: Participants
Arm/Group | Placebo | Active
Number analyzed (Participants) | 11 | 14
Participants
  Positive | 10 | 11
  Negative | 1 | 3
Statistical Analysis 1: Comparison: Placebo vs Active; Test type: Superiority; p = 0.6043, Fisher Exact

17. Secondary Outcome: Detection of Viremia (Blood) by PCR Six Weeks After Trial Entry
Description: Each subject either has positive or negative PCR results. Virus is detected if the PCR is positive.
Time Frame: At 6 weeks (Day 42)
Measure: Number; unit: Participants
Arm/Group | Placebo | Active
Number analyzed (Participants) | 15 | 14
Participants
  Positive | 4 | 2
  Negative | 11 | 12
Statistical Analysis 1: Comparison: Placebo vs Active; Test type: Superiority; p = 0.6513, Fisher Exact

18. Secondary Outcome: Detection of Viremia (Blood) by PCR Six Month After Trial Entry
Description: Each subject either has positive or negative PCR results. Virus is detected if the PCR is positive.
Time Frame: At 6 months
Measure: Number; unit: Participants
Arm/Group | Placebo | Active
Number analyzed (Participants) | 15 | 15
Participants
  Positive | 4 | 3
  Negative | 11 | 12
Statistical Analysis 1: Comparison: Placebo vs Active; Test type: Superiority; p = 1.0, Fisher Exact

19. Secondary Outcome: Detection of CMV in Saliva by PCR Six Weeks After Trial Entry
Description: Each subject either has positive or negative PCR results. Virus is detected if the PCR is positive.
Time Frame: At 6 weeks (Day 42)
Measure: Number; unit: Participants
Arm/Group | Placebo | Active
Number analyzed (Participants) | 16 | 16
Participants
  Positive | 9 | 3
  Negative | 7 | 13
Statistical Analysis 1: Comparison: Placebo vs Active; Test type: Superiority; p = 0.0659, Fisher Exact

20. Secondary Outcome: Detection of CMV in Saliva PCR Six Month After Trial Entry
Description: Each subject either has positive or negative PCR results. Virus is detected if the PCR is positive.
Time Frame: At 6 months
Measure: Number; unit: Participants
Arm/Group | Placebo | Active
Number analyzed (Participants) | 16 | 16
Participants
  Positive | 8 | 7
  Negative | 8 | 9
Statistical Analysis 1: Comparison: Placebo vs Active; Test type: Superiority; p = 1.0, Fisher Exact

21. Secondary Outcome: The Quantitative Log Change in Viremia From Baseline to Month 6.
Description: The quantitative change (Month 6 minus baseline) in viremia (blood) Quantitative viral load by PCR in log 10 units measured in urine after 6 weeks of therapy; if undetectable, viral load is assigned a value of 10 (1 in log 10 units).
Time Frame: Baseline to month 6
Population: Overall number of participants analyzed=34: 17 active and 17 placebo
Measure: Least Squares Mean (95% Confidence Interval); unit: log10 IU/ml
Arm/Group | Randomized Group
Number analyzed (Participants) | 34
log10 IU/ml
  Active: number analyzed (Participants) | 17
  Active | 0.4908 [0.08108 to 0.9005]
  Placebo: number analyzed (Participants) | 17
  Placebo | -0.1528 [-0.5721 to 0.2664]

22. Secondary Outcome: The Quantitative Log Reduction in Viruria Detected After 6 Weeks of Therapy
Description: The quantitative log reduction in viruria (urine) detected after 6 weeks of therapy. Quantitative viral load by PCR in log 10 units measured in urine after 6 weeks of therapy; if undetectable, viral load is assigned a value of 10 (1 in log 10 units)
Time Frame: Baseline thru months 6
Population: Overall number of participants analyzed=28: 15 active and 13 placebo
Measure: Least Squares Mean (95% Confidence Interval); unit: log10 IU/ml
Arm/Group | Randomized Group
Number analyzed (Participants) | 28
log10 IU/ml
  Active: number analyzed (Participants) | 15
  Active | 1.2152 [0.5274 to 1.9029]
  Placebo: number analyzed (Participants) | 13
  Placebo | 0.8390 [-0.05057 to 1.7286]

23. Secondary Outcome: The Quantitative Log Reduction in CMV in Saliva Detected After 6 Weeks of Therapy
Description: The quantitative log reduction in CMV in saliva (urine) detected after 6 weeks of therapy. Quantitative viral load by PCR in log 10 units measured in urine after 6 weeks of therapy; if undetectable, viral load is assigned a value of 10 (1 in log 10 units)
Time Frame: Baseline thru months 6
Population: Overall number of participants analyzed=34
Measure: Least Squares Mean (95% Confidence Interval); unit: log10 IU/ml
Arm/Group | Randomized Group
Number analyzed (Participants) | 34
log10 IU/ml
  Active: number analyzed (Participants) | 17
  Active | 1.3202 [0.6894 to 1.9509]
  Placebo: number analyzed (Participants) | 17
  Placebo | 0.0057 [-0.6395 to 0.6508]

24. Secondary Outcome: Number of Adverse Events in the Active Group That Resulted in Discontinuation of Valganciclovir
Description: AE resulting in discontinuation of valganciclovir (active group only). This outcome summarizes the number of adverse events (AEs) that resulted in the discontinuation of valganciclovir in the active group only.
Time Frame: Day 1 thru day 70
Population: No participants in the active group were discontinued due to adverse event.
Measure: Number; unit: Participants
Groups:
- Randomized Group: Randomized children between 1 month and 3 years of age (up to 4th birthday) with sensoneural hearing loss and documented CMV infection will receive valganciclovir orally twice a day for 6 weeks
Arm/Group | Randomized Group
Number analyzed (Participants) | 17
Participants
  No | 17
  Yes | 0

25. Secondary Outcome: Adverse Event (AE) Resulting in Unresolved Outcome
Description: Adverse event resulting in unresolved outcome. This outcome summarizes the number of adverse events (AEs) that resulted in unresolved outcome of that AE.
Time Frame: Day 1 thru day 70
Population: Overall number of participants analyzed=18
Measure: Number; unit: Participants
Arm/Group | Placebo | Active
Number analyzed (Participants) | 18 | 17
Participants
  No | 18 | 17
  Yes | 0 | 0

26. Secondary Outcome: Adverse Event (AE) Resulting in Unanticipated Medically Attended Visit
Description: Adverse event resulting in unanticipated medically attended visit. This outcome summarizes the number of adverse events (AEs) that resulted in the unanticipated medically attended visit.
Time Frame: Day 1 thru day 70
Population: Overall number of participants analyzed=18
Measure: Number; unit: Participants
Arm/Group | Placebo | Active
Number analyzed (Participants) | 18 | 17
Participants
  No | 15 | 17
  Yes | 3 | 0

ADVERSE EVENTS:
Time Frame: All AEs and SAEs from Study Day 1 through four weeks following the last dose of study drug. All AEs and SAEs will be followed until resolution, even if this extends beyond the study reporting period. Resolution of an AE is defined as the return to pretreatment status or stabilization of the condition with the expectation that it will remain chronic.
Description: Any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of medicinal (investigational) product whether or not considered drug related. The occurrence of an AE may come to the attention of study personnel during study visits and interviews of a study recipient presenting for medical care, or upon review by a study monitor.
Arm/Group | Placebo | Active
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/18 | 1/17
Other Adverse Events (participants affected / at risk) | 18/35 | 17/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=18) | Active (N=17)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=35) | Active (N=35)
Decrease in hemoglobin (Blood and lymphatic system disorders) | 1/18 (1) | 0/17 (0)
Neutropenia (Blood and lymphatic system disorders) | 2/18 (4) | 1/17 (1)
Monocytopenia (Blood and lymphatic system disorders) | 0/18 (0) | 1/17 (1)
Bilateral ear infection (Ear and labyrinth disorders) | 1/18 (1) | 0/17 (0)
Otitis Media (Ear and labyrinth disorders) | 1/18 (1) | 1/17 (1)
Ear Infection (Ear and labyrinth disorders) | 0/18 (0) | 1/17 (1)
Fall on chin (General disorders) | 1/18 (1) | 0/17 (0)
Fever (General disorders) | 3/18 (3) | 1/17 (1)
Hyperkalemia (General disorders) | 0/18 (0) | 1/17 (1)
Long Sighted (General disorders) | 0/18 (0) | 1/17 (1)
Nose Bleed (General disorders) | 1/18 (1) | 0/17 (0)
Pyrexia (General disorders) | 0/18 (0) | 1/17 (1)
Raised Temperature (General disorders) | 1/18 (1) | 0/17 (0)
Constipation (Gastrointestinal disorders) | 2/18 (3) | 1/17 (1)
Diarrhoea (Gastrointestinal disorders) | 0/18 (0) | 1/17 (1)
Emesis (Gastrointestinal disorders) | 0/18 (0) | 1/17 (1)
Gastroenteritis (Gastrointestinal disorders) | 0/18 (0) | 1/17 (1)
Loose stools (Gastrointestinal disorders) | 1/18 (2) | 0/17 (0)
Reduced Appetite (Gastrointestinal disorders) | 0/18 (0) | 1/17 (1)
Reflux (Gastrointestinal disorders) | 0/18 (0) | 1/17 (1)
Teething (Gastrointestinal disorders) | 2/18 (2) | 2/17 (2)
Viral Gastroenteritis (Gastrointestinal disorders) | 0/18 (0) | 1/17 (1)
Vomiting (Gastrointestinal disorders) | 2/18 (5) | 4/17 (4)
Weight Loss (Gastrointestinal disorders) | 0/18 (0) | 1/17 (1)
Chicken Pox (Infections and infestations) | 1/18 (1) | 0/17 (0)
Hand, Foot and Mouth Disease (Infections and infestations) | 1/18 (1) | 1/17 (1)
Infection at Surgical Incision Site (Infections and infestations) | 0/18 (0) | 1/17 (1)
Rhinitis (Infections and infestations) | 1/18 (1) | 0/17 (0)
Tonsillitis (Infections and infestations) | 1/18 (1) | 1/17 (1)
Viral Illness (Infections and infestations) | 2/18 (3) | 1/17 (1)
Head, Eye and Right Arm Injury--Suspected trauma to lacrimal sac. (Injury, poisoning and procedural complications) | 0/18 (0) | 1/17 (1)
Minor Injury--Bruise Right Eye and Cheek and Left Forehead (Injury, poisoning and procedural complications) | 0/18 (0) | 1/17 (1)
Buckle Fracture of Right Tibia and Fibula (Musculoskeletal and connective tissue disorders) | 0/18 (0) | 1/17 (1)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0/18 (0) | 1/17 (1)
Agitation (Psychiatric disorders) | 1/18 (1) | 0/17 (0)
Crying since first dose (Psychiatric disorders) | 1/18 (1) | 0/17 (0)
Fussiness (Psychiatric disorders) | 1/18 (1) | 0/17 (0)
Hallucination-Nightmare (Psychiatric disorders) | 0/18 (0) | 1/17 (1)
Intermittent Hyperactivity (Psychiatric disorders) | 1/18 (1) | 0/17 (0)
Lethargic and Sleeping more than usual (Psychiatric disorders) | 0/18 (0) | 1/17 (1)
Screaming--Unsettled (Psychiatric disorders) | 0/18 (0) | 1/17 (1)
Blood in Urine (Renal and urinary disorders) | 0/18 (0) | 1/17 (1)
Protein in Urine (Renal and urinary disorders) | 0/18 (0) | 1/17 (1)
Urinary Incontinence (Renal and urinary disorders) | 1/18 (1) | 0/17 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0/18 (0) | 1/17 (1)
Blocked Nose (Respiratory, thoracic and mediastinal disorders) | 0/18 (0) | 1/17 (1)
Bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 0/18 (0) | 2/17 (2)
Coryzal Symptoms (Respiratory, thoracic and mediastinal disorders) | 1/18 (2) | 2/17 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2/18 (5) | 1/17 (1)
Cough and Runny Nose (Respiratory, thoracic and mediastinal disorders) | 0/18 (0) | 1/17 (1)
Cough and Cold (Respiratory, thoracic and mediastinal disorders) | 1/18 (1) | 0/17 (0)
Exacerbation (Respiratory, thoracic and mediastinal disorders) | 0/18 (0) | 1/17 (1)
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 2/18 (2) | 1/17 (1)
Rhinos Virus Infection (Respiratory, thoracic and mediastinal disorders) | 0/18 (0) | 1/17 (1)
Runny Nose (Respiratory, thoracic and mediastinal disorders) | 0/18 (0) | 1/17 (1)
Fine Erythematous, raised rash on Chest and Abdomen (Skin and subcutaneous tissue disorders) | 0/18 (0) | 1/17 (1)
Glass in Foot (Skin and subcutaneous tissue disorders) | 0/18 (0) | 1/17 (1)
Impetigo (Skin and subcutaneous tissue disorders) | 0/18 (0) | 1/17 (1)
Rash (Skin and subcutaneous tissue disorders) | 0/18 (0) | 2/17 (4)
White Discolouration of Lips and Throat (Skin and subcutaneous tissue disorders) | 1/18 (1) | 0/17 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-04-28): https://cdn.clinicaltrials.gov/large-docs/69/NCT01649869/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-14): https://cdn.clinicaltrials.gov/large-docs/69/NCT01649869/SAP_001.pdf